CLINICAL TRIAL: NCT07041632
Title: Can Acupuncture Replace Conscious Sedation in In-Vitro-Fertilization Transvginal Oocyte Retrievals?
Brief Title: Pain Relief in Women Undergoing Oocyte Retrieval (OR) With Electro-acupuncture (EA) or Conscious Sedation (CS) in a Single Assisted Reproduction Centre.
Acronym: EA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Acupuncture in IVF; TCMCRG3103002 (Other: Ministry of Health)
Record Dates: First submitted 2025-05-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pain Intensity Assessment
Keywords: acupuncture, oocyte retrieval, sedation
MeSH Terms: interventions — Conscious Sedation

STUDY DESIGN:
Intervention Model Description: randomised control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electro-acupuncture (Active Comparator): Electro-acupunture is compared to Conscious sedation during egg collection in IVF
  Interventions: Other: electro-acupuncture
- Conscious sedation for egg collection (Active Comparator): Conscious sedation is the common analgesia used in egg collection in IVF
  Interventions: Other: Conscious sedation

INTERVENTIONS:
Other: electro-acupuncture — electro-acupuncture for pain relief in egg collection in IVF
  Arms: electro-acupuncture
Other: Conscious sedation — IVf egg collection using conscious sedation as the usual analgesia
  Arms: Conscious sedation for egg collection

SUMMARY:
This study aims to determine whether one can replace pain relief in women undergoing oocyte retrieval (OR) using electro-acupuncture (EA) instead of conscious sedation (CS).

DETAILED DESCRIPTION:
A total of 60 women were randomized and 29 women were on electro-acupuncture (EA) versus 27 women on conscious sedation (CS) with intravenous medication for transvaginal egg extraction (OR) in IVF. Pain scores were recorded before , during and after egg extraction when the women were on conscious sedation and electro-acupuncture. Side effects were recorded. Physical parameters were recorded. Livebirth outcome were also recorded.

ELIGIBILITY:
Inclusion Criteria: all women undergoing ivf and have given consent -

Exclusion Criteria: women who have infectious skin diseases, women who were unwilling to accept acupunture, history of bleeding disorders.

-

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — ivf female patients
Enrollment: 60 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Pain relief during egg collection | from start of egg collection. to 120 minutes after egg collection
  Pain score 1 to 10 during egg collection in IVF compared between using acupuncture and conscious sedation

SECONDARY OUTCOMES:
Stress, satisfaction measurement and physical parameters between acupuncture and conscious sedation during egg collection in IVF | Up to 120 minutes after egg collection
  Stress score and satisfaction outcome scores 0 to 10 for pain relief between acupuncture and conscious sedation during egg collection were recorded. For the stress score, zero is equivalent to no stress and 10 indicates the worst possible stress. For the satisfaction score, zero is equivalent to no satisfaction at all and 10 is the highest satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Su Ling Yu, FRCOG, Principal Investigator
Locations (1):
- Centre for Assisted Reproduction, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
This study has completed a few years ago.